CLINICAL TRIAL: NCT02807363
Title: A Randomized, Open-label, Parallel-group, Active-control PK/PD Study of Three Doses of Leuprolide Oral Tablets in Comparison to an IM Dose of Leuprolide in Healthy Female Volunteers
Brief Title: A Study of Pharmacokinetic/Pharmacodynamic Profile of Orally Administered Leuprolide in Healthy Female Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enteris BioPharma Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOPDT-ENDO-01
Record Dates: First submitted 2016-06-14; First posted 2016-06-21 (Estimated); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Endometriosis
Keywords: endometriosis; gonadotropin-releasing hormone agonist; healthy volunteers; leuprolide oral tablet
MeSH Terms: conditions — Endometriosis | interventions — Leuprolide; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A: Leuprolide Oral Tablet, 4 mg QD (Experimental): Leuprolide Oral Tablet QD: 4 mg for 28 consecutive days.
  Interventions: Drug: Leuprolide Oral Tablet 4-mg QD
- Treatment B: Leuprolide Oral Tablet, 4 mg BID (Experimental): Leuprolide Oral Tablet BID: 4 mg, 12 hours apart for 28 consecutive days.
  Interventions: Drug: Leuprolide Oral Tablet 4-mg BID
- Treatment C: Leuprolide 1 month depot (Active Comparator): Leuprolide Depot : intramuscular (IM) 3.75 mg depot injection administered for one month of therapy
  Interventions: Drug: Leuprolide Depot
- Treatment D: Leuprolide Oral Tablet, 10 mg BID (Experimental): Leuprolide Oral Tablet BID: 10 mg, 12 hours apart for 28 consecutive days
  Interventions: Drug: Leuprolide Oral Tablet 10-mg BID

INTERVENTIONS:
Drug: Leuprolide Oral Tablet 4-mg QD — 4-mg Leuprolide oral tablet once daily for 28 consecutive days.
  Other Names: Ovarest™ 4.0 mg
  Arms: Treatment A: Leuprolide Oral Tablet, 4 mg QD
Drug: Leuprolide Oral Tablet 4-mg BID — 4-mg Leuprolide oral tablet twice daily for 28 consecutive days.
  Other Names: Ovarest™ 4.0 mg
  Arms: Treatment B: Leuprolide Oral Tablet, 4 mg BID
Drug: Leuprolide Depot — 3.75 mg intramuscular depot injection
  Other Names: Lupron Depot® 3.75 mg
  Arms: Treatment C: Leuprolide 1 month depot
Drug: Leuprolide Oral Tablet 10-mg BID — 10-mg Leuprolide oral tablet twice daily for 28 consecutive days.
  Other Names: Ovarest™ 10.0 mg
  Arms: Treatment D: Leuprolide Oral Tablet, 10 mg BID

SUMMARY:
This Phase 2a, pharmacokinetic/pharmacodynamic study will determine the safety and provide evaluation of the PK/PD metrics of three different oral doses selected upon the results of the study LOPDT-PH1-01 - 4 mg oral tablets administered over 28 days as QD and BID regimens and 10 mg oral tablets administered over 28 days as a BID regimen. The PK/PD profiles of the study drug will be compared to the leuprolide formulation approved for the treatment of endometriosis (a monthly intramuscular injection, Lupron Depot 3.75 mg). Major PK (e.g., a total exposure to leuprolide) and PD parameters (e.g., rates of the estradiol suppression and cessation of the menstrual period) will also be evaluated against the Lupron Depot historical data.

DETAILED DESCRIPTION:
Site initiation visit of the study site, InVentiv Health Clinique, Inc. by on-site visit and teleconference was done and the final report signed 21st July 2017.

For the demographic and baseline characteristics descriptive statistics consisting of mean, median, standard deviation, minimum, maximum and sample size is reported for continuous variables like age, body mass index, weight and height. categorical variables like ethnicity, gender and race is presented as frequency counts and percentages.

For PK analysis, Steady state concentration level of leuprolide calculated for oral tablets (Treatments A and B) at the end of the fourth treatment week (Treatment Days 28) as the 24-hour AUCs divided by the duration of the dosing interval i.e., 24 hours.

For PD analysis, subject incidence of estradiol level below 40 pg/mL was assessed. The ovulation rate determined by the extent of progesterone suppression is presented.

Only observed data is used in the data analysis except for concentration values below the lower limit of quantitation (BLQ) and samples with no reportable value occurring prior to dosing (on Day 1 only). No attempt is made to impute (i.e., extrapolate or interpolate) estimates for missing data.

For safety analysis, incidence of treatment emergent adverse events both during the dosing and post dosing period is presented.

The Medical Dictionary for Regulatory Activities (MedDRA®) Version 20.1 is used to classify all medical history findings and incidences of treatment emergent adverse events (TEAE) reported during the study by System Organ Class (SOC) and Preferred Term (PT).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy premenopausal female volunteers, aged 18 to 49 years;
2. Body mass index (BMI) ≥ 18 and ≤ 32 kg/m2, and weight ≥ 110 lb (approximately 50 kg);
3. Regular menstrual cycles with a usual length ranging from 21 days to 35 days. If subject had recently used hormonal birth control, historical data prior to use were used to determine qualification and must also meet this criterion;
4. If of childbearing potential and sexually active with a risk of pregnancy, willing to use one of the following acceptable methods of contraception throughout the study and for at least 30 days after the last drug administration:

   1. intrauterine contraceptive device (IUD) without hormone release system placed at least 4 weeks prior to the first study drug administration with simultaneous use of condom for the male partner;
   2. simultaneous use of diaphragm with intravaginally applied spermicide and condom for the male partner starting at least 14 days prior to drug administration;
   3. sterile male partner (vasectomized for at least 6 months); Note: Surgically sterile subjects who have had a tubal ligation were considered of non-childbearing potential and were not required to use contraception;
5. Willing to refrain from excessive use of alcohol during the entire study and willing to refrain from use of alcohol 24 hours prior to any PK blood draw taken during the study;
6. Willing to refrain from use of prescription medications, over-the-counter medications, and natural health products during the entire study;
7. Willing and capable to give informed consent to participate in study.

Exclusion Criteria:

1. Hypersensitivity to GnRH, GnRH agonist analogs, similar nonapeptides, or any of the excipients in Lupron Depot®. Note: This was a contraindication from the Lupron Depot® label;
2. Undiagnosed abnormal vaginal bleeding. Note: This was a contraindication from the Lupron Depot® label;
3. Known or suspected pregnancy, or subjects who were considered to become pregnant prior to the conclusion of this study. Note: Lupron Depot® was contraindicated in women who were or may become pregnant while receiving the drug. Lupron Depot® could cause fetal harm when administered to a pregnant woman. If this drug was used during pregnancy, or if the patient becomes pregnant while taking this drug, the patient should be apprised of the potential hazard to the fetus;
4. Breastfeeding or within 2 months after stopping breastfeeding (relative to the Screening visit). Note: Use of Lupron Depot® was contraindicated in women who were breastfeeding;
5. Thrombophlebitis, thromboembolic disorders, cerebral apoplexy, or a past history of these conditions. Note: Per the Lupron Depot® label, a possible coadministration of norethindrone acetate was contraindicated in women with thrombophlebitis, thromboembolic disorders, cerebral apoplexy, or a past history of these conditions
6. Markedly impaired liver function or liver disease. Note: Per the Lupron Depot® label, a possible co-administration of norethindrone acetate was contraindicated in women with markedly impaired liver function or liver disease;
7. Known or suspected carcinoma of the breast. Note: Per the Lupron Depot® label, a possible co-administration of norethindrone acetate was contraindicated in women with known or suspected carcinoma of the breast;
8. Status postpartum or post-abortion within a period of 2 months prior to the Screening visit;
9. A cervical cytology smear of Papanicolaou (Pap) Class III or greater or a Bethesda System report of low grade squamous intraepithelial lesions (SIL) or greater (Pap smear results within last 12 months were acceptable if properly documented);
10. Use of any tobacco products (including electronic cigarettes) in the 3 months preceding the Screening visit or positive urine cotinine test at Screening;
11. History of significant alcohol or drug abuse within 1 year prior to the Screening visit;
12. Clinically significant (CS) vital sign abnormalities (systolic blood pressure [BP] lower than 90 or over 140 mm Hg, diastolic BP lower than 50 or over 90 mm Hg, or heart rate less than 50 or over 100 bpm) at Screening;
13. Any CS history or presence of neurologic, endocrinologic, pulmonary, hematologic, immunologic, or metabolic disease;
14. History of severe respiratory depression or pulmonary insufficiency;
15. Diabetes mellitus requiring insulin;
16. History of headaches with focal neurological symptoms;
17. Uncontrolled thyroid disorder;
18. Sickle cell anemia;
19. Current or history of CS depression in the last year;
20. Known disturbance of lipid metabolism;
21. Hepatic adenoma or carcinoma;
22. Known or suspected endometrial carcinoma or estrogen-dependent neoplasia;
23. Clinically significant history or presence of any gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting) or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug;
24. Difficulty in swallowing study medication;
25. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Investigator, could contraindicate the subject's participation in this study;
26. Positive test for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) at Screening;
27. Administration of any investigational drug and/or experimental device within 30 days prior to the Screening visit;
28. Administration of any biologics within 90 days prior to the Screening visit;
29. Clinically significant finding on the electrocardiogram (ECG) suggesting participation in the study could pose a risk to the subject;
30. A depot injection or an implant of any drug within 6 months prior to the Screening visit;
31. Use of oral contraceptives or other sex steroid hormones within 3 months prior to the Screening visit;
32. Any CS physical or gynecological abnormality at the Screening visit;
33. Any CS abnormal laboratory test result at the Screening visit;
34. Hemoglobin < 115 g/L and/or hematocrit < 0.32 L/L;
35. Use of prescription medication within 14 days prior to the first administration of study medication or over-the-counter (OTC) products (including natural health products; e.g., food supplements, vitamins, herbal supplements) within 7 days prior to the first administration of study medication, except for topical products without significant systemic absorption;
36. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at Screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing;
37. Deemed by the Investigator to have questionable ability to comply with the study protocol;
38. History of seizures, epilepsy, cerebrovascular disorders, central nervous system (CNS) anomalies or tumors;
39. Significant risk factors for decreased bone mineral content and/or bone mass, such as family history (in a first degree relative) of osteoporosis, personal history of chronic use of corticosteroids or anticonvulsants.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pre-menopausal female volunteers
Enrollment: 35 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Shangold, MD, Study Chair — Enteris BioPharma Inc.
Locations (1):
- inVentiv Health Clinique, Inc., Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Leuprolide Oral Tablet, 4 mg QD (Treatment A): Leuprolide Oral Tablet QD: 4 mg for 28 consecutive days.
  Leuprolide Oral Tablet 4-mg QD: 4-mg Leuprolide oral tablet once daily for 28 consecutive days.
- Leuprolide Oral Tablet, 4 mg BID (Treatment B): Leuprolide Oral Tablet BID: 4 mg, 12 hours apart for 28 consecutive days.
  Leuprolide Oral Tablet 4-mg BID: 4-mg oral tablet twice daily for 28 consecutive days.
- Leuprolide 1 Month Depot (Treatment C): Leuprolide Depot : intramuscular (IM) 3.75 mg depot injection administered for one month of therapy
  Leuprolide Depot: 3.75 mg intramuscular depot injection
- Leuprolide Oral Tablet, 10 mg BID (Treatment D): Leuprolide Oral Tablet BID: 10 mg, 12 hours apart for 28 consecutive days
  Leuprolide Oral Tablet 10-mg BID: 10-mg oral tablet twice daily for 28 consecutive days.
Period: Dosing Period
Arm/Group | Leuprolide Oral Tablet, 4 mg QD (Treatment A) | Leuprolide Oral Tablet, 4 mg BID (Treatment B) | Leuprolide 1 Month Depot (Treatment C) | Leuprolide Oral Tablet, 10 mg BID (Treatment D)
Started | 9 | 9 | 5 | 12
Completed | 9 | 8 | 5 | 12
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Post- Dosing Period
Arm/Group | Leuprolide Oral Tablet, 4 mg QD (Treatment A) | Leuprolide Oral Tablet, 4 mg BID (Treatment B) | Leuprolide 1 Month Depot (Treatment C) | Leuprolide Oral Tablet, 10 mg BID (Treatment D)
Started | 9 | 8 | 5 | 12
Completed | 9 | 8 | 5 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leuprolide Oral Tablet, 4 mg QD (Treatment A) | Leuprolide Oral Tablet, 4 mg BID (Treatment B) | Leuprolide 1 Month Depot (Treatment C) | Leuprolide Oral Tablet, 10 mg BID (Treatment D) | Total
Number analyzed (Participants) | 9 | 9 | 5 | 12 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (6.1) | 38.4 (5.9) | 37.8 (6.6) | 37.2 (4.9) | 37.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 5 | 12 | 35
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 1 | 1 | 5
  Not Hispanic or Latino | 6 | 9 | 4 | 11 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 3
  White | 8 | 9 | 5 | 10 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: inches] | 63.93 (2.14) | 63.60 (1.10) | 65.28 (2.69) | 64.05 (2.15) | 64.1 (2.0)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.734 (3.292) | 26.054 (3.262) | 24.242 (3.255) | 24.988 (3.235) | 25.3 (3.2)
Weight [Mean (Standard Deviation); unit: lbs] | 149.41 (22.36) | 149.63 (20.63) | 147.40 (17.47) | 146.64 (22.38) | 148.15 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adequacy of Suppression of Estradiol (E2) as Assessed by Estradiol Level Below 40 pg/mL
Description: Criterion: E2 level is considered suppressed during the evaluation period if a value below pre-specified threshold was reported at least once during that period.
  The days in the row title indicate the evaluation interval.
Time Frame: Dosing Period: Day 8 to 28, Post-dosing: Day 1 to day 28 of post dosing period; Day 29 is the post dosing day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Leuprolide Oral Tablet, 4 mg QD (Treatment A) | Leuprolide Oral Tablet, 4 mg BID (Treatment B) | Leuprolide 1 Month Depot (Treatment C) | Leuprolide Oral Tablet, 10 mg BID (Treatment D)
Number analyzed (Participants) | 9 | 8 | 5 | 12
Participants
  Days 8,15, 22, 28 and 29 | 6 | 7 | 5 | 12
  Days 15, 22, 28 and 29 | 5 | 7 | 5 | 12
  Days 22, 28 and 29 | 4 | 6 | 5 | 9
  Days 22 and 29 | 4 | 6 | 5 | 9
  Entire 28-day Dosing Period | 7 | 8 | 5 | 12
  28-day Post-dosing Period | 7 | 6 | 5 | 9

2. Primary Outcome: Ovulation Rate - Measured by Number of Subjects With Progesterone Levels Not Less Than 3000 pg/mL
Description: Progesterone level is considered suppressed during the evaluation period if a value below pre-specified threshold (3000 pg/mL) was reported at least once during that period.
  The days in row title indicate the evaluation interval.
Time Frame: Dosing period: Day 1 to Day 28 and 28 day Post-Dosing Period; 29 day is post dosing day 1
Measure: Count of Participants; unit: Participants
Groups:
- Leuprolide 1 Month Depot (Treatment C): Leuprolide Depot : intramuscular (IM) 3.75 mg depot injection administered for one month (28 day cycle) of therapy
  Leuprolide Depot: 3.75 mg intramuscular depot injection
Arm/Group | Leuprolide Oral Tablet, 4 mg QD (Treatment A) | Leuprolide Oral Tablet, 4 mg BID (Treatment B) | Leuprolide 1 Month Depot (Treatment C) | Leuprolide Oral Tablet, 10 mg BID (Treatment D)
Number analyzed (Participants) | 9 | 8 | 5 | 12
Participants
  Days 8, 15, 22, 28 and 29 | 4 | 3 | 3 | 10
  Days 15, 22, 28 and 29 | 2 | 2 | 0 | 0
  Days 22, 28 and 29 | 2 | 2 | 0 | 0
  Days 22 and 29 | 2 | 1 | 0 | 0
  Entire 28-day Dosing Period | 8 | 5 | 4 | 12
  28-day Post-dosing Period | 9 | 7 | 2 | 12

3. Primary Outcome: Number of Subjects Who Experienced Treatment Emergent Adverse Events (TEAE) Excluding Menstrual Disorders
Description: The participant incidence of TEAEs was generally comparable during the dosing period across the treatment groups.
  Treatment C is a depot formulation established to release the drug over a period of 1 month. The data for adverse event was collected for day 1 to 28 of the dosing period.
Time Frame: Dosing Period: Day 1 to day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Leuprolide Oral Tablet, 4 mg QD (Treatment A) | Leuprolide Oral Tablet, 4 mg BID (Treatment B) | Leuprolide 1 Month Depot (Treatment C) | Leuprolide Oral Tablet, 10 mg BID (Treatment D)
Number analyzed (Participants) | 9 | 9 | 5 | 12
Participants
  Number of subjects with at least one TEAE | 7 | 9 | 4 | 8
  Number of subjects who discontinued due to TEAE | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Subjects Who Experienced Treatment-Emergent Adverse Events (TEAEs), Excluding Menstrual Disorders
Description: Treatment C is a depot formulation established to release the drug over a period of 1 month. The data for post dosing adverse event was collected starting from day 1 to 28 post the 28th day of dosing.
Time Frame: Post dosing period (starting day 1 to day 28 post dosing period)
Measure: Count of Participants; unit: Participants
Groups:
- Leuprolide 1 Month Depot(Treatment C): Leuprolide Depot : intramuscular (IM) 3.75 mg depot injection administered for one month of therapy
  Leuprolide Depot: 3.75 mg intramuscular depot injection
Arm/Group | Leuprolide Oral Tablet, 4 mg QD (Treatment A) | Leuprolide Oral Tablet, 4 mg BID (Treatment B) | Leuprolide 1 Month Depot(Treatment C) | Leuprolide Oral Tablet, 10 mg BID (Treatment D)
Number analyzed (Participants) | 9 | 8 | 5 | 12
Participants
  Number of subjects with at least one TEAE | 1 | 2 | 1 | 3
  Number of subject who discontinued due to TEAEs | 0 | 0 | 0 | 0

5. Primary Outcome: Steady State Concentration Level, (Css) of Leuprolide
Description: Treatment A and B: Steady state concentration level calculated for oral tablets at the end of the fourth treatment week (Treatment Day 28) as the 24-hour AUCs divided by the duration of the dosing interval i.e. 24 hours.
  Treatment C: Steady state concentration level calculated for IM injection at the fourth treatment week (a mean of leuprolide levels on Days 22 and 29).
Time Frame: Treatment Day 28 for oral groups; Treatment Days 22-29 for Lupron Depot group
Population: Treatment D: Css determination along with most other pharmacokinetic parameters was not done for this treatment arm as fewer blood samples were planned for this treatment arm.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Leuprolide Oral Tablet, 4 mg QD (Treatment A) | Leuprolide Oral Tablet, 4 mg BID (Treatment B) | Leuprolide 1 Month Depot (Treatment C) | Leuprolide Oral Tablet, 10 mg BID (Treatment D)
Number analyzed (Participants) | 8 | 8 | 5 | 0
pg/mL | 357.80 (367.37) | 688.27 (258.01) | 180.95 (101.04) |

ADVERSE EVENTS:
Time Frame: Dosing period (day 1 to day 28) and post dosing period (day 1 to day 28)
Description: Treatment C being a 1 month (28 day cycle) depot formulation is mentioned as a 1 month therapy but the adverse event monitoring was done for the same time frame as treatment A, B and D.
Arm/Group | Leuprolide Oral Tablet, 4 mg QD (Treatment A) | Leuprolide Oral Tablet, 4 mg BID (Treatment B) | Leuprolide 1 Month Depot (Treatment C) | Leuprolide Oral Tablet, 10 mg BID (Treatment D)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/5 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/5 | 0/12
Other Adverse Events (participants affected / at risk) | 7/9 | 9/9 | 4/5 | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprolide Oral Tablet, 4 mg QD (Treatment A) (N=9) | Leuprolide Oral Tablet, 4 mg BID (Treatment B) (N=9) | Leuprolide 1 Month Depot (Treatment C) (N=5) | Leuprolide Oral Tablet, 10 mg BID (Treatment D) (N=12)
Headache, disturbance in attention, dizziness, presyncope (Nervous system disorders) | 4 (6) | 8 (10) | 3 (3) | 4 (4)
Nausea, Vomiting, Abdominal pain, abdominal pain upper, dry mouth, faeces soft (Gastrointestinal disorders) | 0 (0) | 5 (6) | 1 (2) | 2 (5)
hot flush (Vascular disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (4)
Breast tenderness. Metrorrhagia, (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Acne, erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Nasopharyngitis, gastroenteritis, vaginitis gardnerella (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cough, Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Depressed mood, Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02807363/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT02807363/SAP_001.pdf